CLINICAL TRIAL: NCT06156709
Title: The Effect of Using Local Anesthetics in a Higher Volume and Lower Dose On Analgesic Quality of Labor Analgesia With Dural Puncture Epidural Technique: Double-Blind Randomised Controlled Study
Brief Title: Effect of Higher Volume and Lower Dose on Analgesic Quality During Labor Analgesia With Dural Puncture Epidural
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Clinical Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/829
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): The patients will be given 10 ml of a solution containing 0,1% of bupivacaine and 2 mcg/ml fentanyl through the epidural cathether. Level of sensory block will be tested by testing with ice from S2 dermatome cephally.
  Analgesia will be maintained by programmed intermittant epidural (PIE) boluses of 7,5 ml of the same solution once in every hour, starting 1 hour after the loading dose. In addition, patient controlled epidural analgesia (PCEA) will be programmed so that 8 ml of the same solution with a lock-time of 10 ml may be administered. "Breakthrough pain" that requires even further analgesia will be treated with an epidural bolus of 5 ml of 0,125% bupivacain solution.
  Interventions: Procedure: Group I: Lower Volume with Higher Anaesthetic Concentration
- Group II (Active Comparator): The patients will be given 20 ml of a solution containing 0,0625% of bupivacaine and 2 mcg/ml fentanyl through the epidural cathether. Analgesia will be maintained by programmed intermittant epidural boluses of 15 ml of the same solution once in every hour, starting 1 hour after the loading dose. In addition, patient controlled epidural analgesia (PCEA) will be programmed so that 8 ml of the same solution with a lock-time of 10 ml may be administered. "Breakthrough pain" that requires even further analgesia will be treated with an epidural bolus of 5 ml of 0,125% bupivacain solution.
  Interventions: Procedure: Group II: Higher Volume with LowerAnaesthetic Concentration

INTERVENTIONS:
Procedure: Group I: Lower Volume with Higher Anaesthetic Concentration — 10 ml of a solution containing 0,1% of bupivacaine and 2 mcg/ml fentanyl through the epidural cathether, maintained by programmed intermittant epidural (PIE) boluses of 7,5 ml of the same solution once in every hour, starting 1 hour after the loading dose. patient controlled epidural analgesia (PCEA) will be programmed so that 8 ml of the same solution with a lock-time of 10 ml may be administered
  Arms: Group I
Procedure: Group II: Higher Volume with LowerAnaesthetic Concentration — 20 ml of a solution containing 0,0625% of bupivacaine and 2 mcg/ml fentanyl through the epidural cathether, maintained by programmed intermittant epidural boluses of 15 ml of the same solution once in every hour, starting 1 hour after the loading dose. patient controlled epidural analgesia (PCEA) will be programmed so that 8 ml of the same solution with a lock-time of 10 ml may be administered
  Arms: Group II

SUMMARY:
It is aimed in this study to compare the effect of using local anaesthetics in a higher volume and lower dose on the total anesthetic consumption and quality of labor analgesia with dural puncture epidural technique.

DETAILED DESCRIPTION:
This study will be conducted as a prospective randomized, controlled, double-blind trial following the approval of the ethical committee at Atatürk University Medical Faculty Hospital and after obtaining written consent from the participating patients. The study will include pregnant women aged 20 to 45 with American Society of Anesthesiologists (ASA) II classification, full-term, nulliparous and singleton pregnancies. Using a randomisation procedure, the participants will be allocated into two equal groups: Group I and Group II.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy nulliparous women
2. American Society of Anaesthesiology Score of II
3. During active labor
4. At weeks 37-42.
5. Singlet vertex presentation
6. Cervical dilation <5 cm at the request of labor analgesia
7. VAS score >40

Exclusion Criteria:

1. Age <20 or >45,
2. Morbid obesity
3. Presence of pregnancy-related comorbidities (e.g: gestational diebetes, gestational hypertension and preeclampsia)
4. History of drug abuse
5. Contrindication for neuraxial blocks
6. Conditions that increase the risk of need for cesarean section (e.g. placenta previa, uterus abnormalities or surgeries)
7. Diagnosed fetal abnormalities
8. Cases where dura gets punctured unintendedly with the epiduralneedle
9. Cases where flow of cerebrospinal fluid (CSF) is not observed after dural puncture
10. Cases where a cesarean section is performed at any stage of labor
11. Cases where labor is completed in 1 hour from the start of analgesia procedure.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference between total local anaesthetic consumption | 5 hours or before if the labor is completed
  The study will involve monitoring the patients starting 2 minutes after the initial epidural dose, every 2 minutes during the first 20 minutes. Monitoring will continue at the 30th minute, and once in every 90 minutes for 5 hours or until labor is completed.
  Total bupivacain consumption will be calculated as follows: PIEB + PCEA + boluses by the clinician. Bupivacain consumption per hour will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Dostbil, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Suzuki N, Koganemaru M, Onizuka S, Takasaki M. Dural puncture with a 26-gauge spinal needle affects spread of epidural anesthesia. Anesth Analg. 1996 May;82(5):1040-2. doi: 10.1097/00000539-199605000-00028. PMID 8610864
- [Background] Thomas JA, Pan PH, Harris LC, Owen MD, D'Angelo R. Dural puncture with a 27-gauge Whitacre needle as part of a combined spinal-epidural technique does not improve labor epidural catheter function. Anesthesiology. 2005 Nov;103(5):1046-51. doi: 10.1097/00000542-200511000-00019. PMID 16249679
- [Background] Wilson SH, Wolf BJ, Bingham K, Scotland QS, Fox JM, Woltz EM, Hebbar L. Labor Analgesia Onset With Dural Puncture Epidural Versus Traditional Epidural Using a 26-Gauge Whitacre Needle and 0.125% Bupivacaine Bolus: A Randomized Clinical Trial. Anesth Analg. 2018 Feb;126(2):545-551. doi: 10.1213/ANE.0000000000002129. PMID 28622178
- [Background] Kaddoum R, Motlani F, Kaddoum RN, Srirajakalidindi A, Gupta D, Soskin V. Accidental dural puncture, postdural puncture headache, intrathecal catheters, and epidural blood patch: revisiting the old nemesis. J Anesth. 2014 Aug;28(4):628-30. doi: 10.1007/s00540-013-1761-y. Epub 2013 Dec 18. PMID 24347033